CLINICAL TRIAL: NCT06643689
Title: Tranilast Vs. Steroids to Prevent Esophageal Stricture (TAPES) Following Circumferential Endoscopic Submucosal Dissection (cESD) for Superficial Neoplasms
Brief Title: Tranilast Vs. Steroids to Prevent Esophageal Stricture (TAPES) After Endoscopic Resection for Superficial Neoplasms
Acronym: TAPES
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The Third People's Hospital of Hangzhou (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-1044
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Esophageal Stricture; Esophageal Neoplasms
Keywords: Tranilast; Esophageal Neoplasms; Steroids; Esophageal stricture; Circumferential Endoscopic Submucosal Dissection
MeSH Terms: conditions — Esophageal Stenosis; Esophageal Neoplasms | interventions — tranilast; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel groups (Tranilast group and steroid group). Each group will receive their respective treatments concurrently, and outcomes will be assessed independently for each group. This model ensures that participants are not crossed over between treatment arms during the study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single-Blind Method with Investigator Blinding
  Specific blinding measures:
  1. Randomization and drug allocation: Randomization and drug allocation should be managed by a third party (e.g., data management team or pharmacist). The treatment options (Tranilast or steroids) should be distributed in identical appearance, packaging, and dosage forms to ensure that the investigators cannot determine the group assignment based on the drug's appearance.
  2. Protection of subject information: Ensure that investigators have no access to any information regarding the drug name and group assignment. Anonymous numbers or subject codes can be used for labeling, with only the personnel or system responsible for drug allocation knowing the specific group assignments.
  3. Data monitors or independent assessors: Independent monitors or assessors can be introduced, responsible only for follow-up and evaluation of post-procedure stricture, without knowledge of the patients' treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranilast Treatment Group (Experimental): Participants in this group will receive Tranilast for the prevention of stricture after cESD of superficial esophageal tumors.
  Interventions: Drug: Tranilast
- Steroid Treatment Group (Active Comparator): Participants in this group will receive steroids for the prevention of stricture after cESD of superficial esophageal tumors.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Tranilast — Tranilast is an anti-allergic agent that is hypothesized to prevent stricture formation in patients undergoing cESD for superficial esophageal tumors. Participants in this group will receive 100 mg orally three times a day for 8 weeks.
  Arms: Tranilast Treatment Group
Drug: Dexamethasone — Prednisone is a corticosteroid used to reduce inflammation and prevent stricture in patients undergoing cESD for superficial esophageal tumors. Participants in this group will receive an oral dose of 30 mg once daily for 8 weeks, with a gradual tapering of the dosage as follows: Weeks 1-2: 30 mg daily; Weeks 3-4: 25 mg daily; Weeks 5-6: 20 mg daily; Weeks 7-8: 15 mg daily; and then tapering to 10 mg daily in Week 7 and 5 mg daily in Week 8.
  Arms: Steroid Treatment Group

SUMMARY:
The goal of this clinical trial is to learn if tranilast works to prevent esophageal stricture after circumferential endoscopic submucosal dissection (cESD) in adults. It will also help us learn more about the safety of tranilast. The main questions it aims to answer are: 1. Does tranilast reduce the occurence of esophageal stricture in participants after cESD? 2. What medical problems do participants have when taking tranilast.

Researchers will compare tranilast to prednisone (a steroid used in clinical practice with potential defects) to see if tranilast works well to prevent esophageal stricture.

Participants will: 1. Take tranilast or prednisone every day for 8 weeks. 2. Attend visit (at clinic or phone) once every 2 weeks for checkups and tests until 16 weeks. 3. Keep a diary of their symptoms and let researchers know during the 16 weeks follow up.

DETAILED DESCRIPTION:
Esophageal strictures are a frequent complication after cESD for superficial esophageal tumors, which significantly affects patients' quality of life and often necessitates repeated endoscopic interventions. Currently, steroids are widely used to prevent post-cESD strictures, but their side effects, including increased risks of infection and delayed wound healing, limit their use. Tranilast, an anti-inflammatory and antifibrotic agent, has shown potential in preventing fibrosis in preclinical studies, but its clinical efficacy in preventing esophageal stricture after cESD remains unclear.

This randomized, parallel, single-blinded non-inferiority trial aims to compare the efficacy and safety of tranilast with steroids in preventing esophageal strictures post-cESD. The primary outcome is the incidence of esophageal stricture within 16 weeks after cESD. It is a composite outcome defined as the inability to pass a standard endoscope (diameter 10.8 mm) through the stricture site at 16 weeks, or the presence of clinical symptoms of esophageal stricture (such as difficulty swallowing solid food) occurring before the endoscopic assessment at 16 weeks. Secondary outcomes include drug-related side effects, postoperative adverse events, and quality of life scores. This study will provide valuable insights into whether tranilast can serve as an effective and safer alternative to corticosteroids in this setting.

ELIGIBILITY:
Inclusion Criteria:

1. age>18 and proficient in Mandarin.
2. underwent cESD treatment for superficial esophageal neoplasms.
3. agree to sign an informed consent form.

Exclusion Criteria:

1. allergic to tranilast.
2. with severe comorbid conditions.
3. pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of esophageal stricture within 16 weeks after cESD | 16 weeks
  a composite outcome defined as the inability to pass a standard endoscope (diameter 10.8 mm) through the stricture site, or the presence of clinical symptoms of esophageal stricture, such as difficulty swallowing solid food, occurring before the endoscopic assessment at 16 weeks.

SECONDARY OUTCOMES:
drug-related side effects | up to 16 weeks
  Occurrence of side effects directly related to tranilast or steroid treatment, as assessed by clinical monitoring and patient reports. These may include gastrointestinal discomfort, allergic reactions, infection, hepatic and renal function impairment, or other systemic effects.
postoperative adverse events | up to 16 weeks
  Occurrence of any adverse events post-surgery, including bleeding, infection, perforation, or other complications. Events will be documented and classified according to the Common Terminology Criteria for Adverse Events.
quality of life score EQ-5D | 16 weeks
  Assess change in Quality of Life (QoL) Score. Patient-reported quality of life, measured using a validated QoL questionnaire to assess the impact of treatment on daily functioning and well-being. Changes in QoL score from baseline to 16 weeks post-treatment will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Yue Yu, Dr., Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (3):
- China (3):
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Shaoxing Central Hospital, Shaoxing, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding the sharing of individual participant data is currently pending further assessment of data protection laws and privacy concerns. We are also awaiting approval from the ethics committee before making a final decision.